CLINICAL TRIAL: NCT05188300
Title: Free Style Pedicled Perforators Propellers Flaps for Meningomylocele Defects Reconstruction With Sequential Advance in Perforators Dissection
Brief Title: Propellers Flaps for Meningomylocele Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel-Tawab Mohamed, Lecturer, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: propellers flap
Record Dates: First submitted 2021-12-26; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Meningocele; Meningomyelocele
Keywords: Reconstructive Surgical Procedures / adverse effects; Meningomyelocele / surgery
MeSH Terms: conditions — Meningocele; Meningomyelocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dorsal intercostal artery (DICA) perforator flaps (Experimental): Retrograde dissection of free style perforator arising from DICA according to region of dorsal spine and identification of paraspinal muscle where perforator vessel was found
  Interventions: Procedure: Freestyle pedicled perforators propellers flaps for meningomyelocele defects
- Trapezius musculocutaneous perforator flaps (Experimental): Retrograde dissection of a free style perforator arising as a trapezius myocutenous perforator where the trapezius muscle is identified and a perforator vessel was isolated.
  Interventions: Procedure: Freestyle pedicled perforators propellers flaps for meningomyelocele defects
- Lumbar artery perforators flaps (Experimental): Retrograde dissection of free style perforator arising from lumbar artery according to region of lumbar spine and identification of lumbar fascia where perforator vessel was found
  Interventions: Procedure: Freestyle pedicled perforators propellers flaps for meningomyelocele defects

INTERVENTIONS:
Procedure: Freestyle pedicled perforators propellers flaps for meningomyelocele defects — Freestyle pedicled perforators propellers flaps for meningomyelocele defects reconstruction with sequential advance in perforators dissection, large number cases, and detailed successful technique.

SUMMARY:
To evaluate reliability of free style propeller perforator flap for coverage MMC soft tissue defect follow a well-established step that overcome the usual problem of pedicled perforators propellers flaps.

DETAILED DESCRIPTION:
Meningomyelocele is a serious congenital birth defect that not only affect mortality and morbidity of neonate but also a lifelong health problem.

The estimated incidence of spina bifida is 1-2 cases per 1000 population. Meningomylocele soft tissue defect reconstruction is considered a lifesaving procedure , the ideal coverage technique should be time limited , reliable and allow healing line to be away from repair of the dura . all of these criteria are available in the selection of free style propeller perforator flap as a method of reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* All cases with dorsolumbar meningomyelocele and age up to 6 months

Exclusion Criteria:

* Infants older than 6 months
* concomitant congenital anomalies
* concomitant spinal kyphosis

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of reconstruction technique | Time of procedure
  Measure the average operative time in minutes in each arm.
Pedicle dissection beyond the muscle | Time of procedure
  Compare the number of pedicle dissection beyond the muscle in each group.

SECONDARY OUTCOMES:
Meningomyelocele Repair Dehiscence and/or CSF leak | Time of procedure
  Compare the number of each complication in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed K Kamel, Principal Investigator — Assiut University; Awni M Shawkat, MD, Study Chair — Assiut University; Mahmoud A Mohamed, Study Director — Assiut University
Locations (1):
- Mohamed Abdeltawab, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kushida-Contreras BH, Gaxiola-Garcia MA. Myelomeningocele defect reconstruction with keystone flaps: vascular rationale for the design and operative technique. Arch Plast Surg. 2021 May;48(3):254-260. doi: 10.5999/aps.2020.01746. Epub 2021 May 15. PMID 34024069
- [Background] Formentin C, de Andrade EJ, Matias LG, Joaquim AF, Tedeschi H, Raposo-Amaral CE, Ghizoni E. Using the keystone design perforator island flap in large myelomeningocele closure. Neurosurg Focus. 2019 Oct 1;47(4):E19. doi: 10.3171/2019.7.FOCUS19383. PMID 31574473
- [Background] Kesan K, Kothari P, Gupta R, Gupta A, Karkera P, Ranjan R, Mutkhedkar K, Sandlas G. Closure of large meningomyelocele wound defects with subcutaneous based pedicle flap with bilateral V-Y advancement: our experience and review of literature. Eur J Pediatr Surg. 2015 Apr;25(2):189-94. doi: 10.1055/s-0034-1368796. Epub 2014 Mar 28. PMID 24683103